CLINICAL TRIAL: NCT05523674
Title: Effects of Warm-up Intensity and Blood Flow Restriction: A Randomized Controlled Clinical Trial
Brief Title: Effects of Warm-up Intensity and Blood Flow Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, Phd Assistant Professor, Paulista University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Warm-up_BRF_FCT/UNESP
Record Dates: First submitted 2022-08-11; First posted 2022-08-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Healthy Men
Keywords: Vascular occlusion; Performance; Body temperature; warm-up
MeSH Terms: interventions — Warm-Up Exercise; Exercise; Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- warm-up performed at 30% VO2max (Experimental): The warm-up exercise will be performed on an ergometric treadmill, through a protocol of 15 minutes duration, with the first 5 minutes of acceleration, until reaching 30% of VO2max, the following 5 minutes of maintenance and the remaining 5 minutes being of slowdown.
  Interventions: Other: Warm-up exercise
- warm-up performed at 80% VO2max (Experimental): The warm-up exercise will be performed on an ergometric treadmill, through a protocol of 15 minutes duration, with the first 5 minutes of acceleration, until reaching 80% of VO2max, the following 5 minutes of maintenance and the remaining 5 minutes being of slowdown.
  Interventions: Other: Warm-up exercise
- warm-up performed at 30% VO2max with Blood Flow Restriction (Experimental): The warm-up exercise will be performed on an ergometric treadmill, through a protocol of 15 minutes of duration, with the first 5 minutes of acceleration, until reaching 30% of VO2max, the following 5 minutes of maintenance and the remaining 5 minutes being of slowdown. During the warm-up exercise, a pressure cuff will be used on each leg, with the blood flow restriction technique (80% of arterial occlusion pressure).
  Interventions: Other: Warm-up exercise with Blood Flow Restriction

INTERVENTIONS:
Other: Warm-up exercise — The warm-up exercise will be performed on a treadmill.
  Other Names: Warming-up; Aerobic Exercise
  Arms: warm-up performed at 30% VO2max; warm-up performed at 80% VO2max
Other: Warm-up exercise with Blood Flow Restriction — The warm-up exercise will be performed on a treadmill and pressure cuffs will be used for the blood flow restriction technique.
  Other Names: Warming-up; Aerobic Exercise; Blood Flow Restriction
  Arms: warm-up performed at 30% VO2max with Blood Flow Restriction

SUMMARY:
Introduction: warming up has the function of preparing the body structures for a given task to be performed during sports, increasing body and muscle temperature, focusing on improving performance. Therefore, the use of the blood flow restriction technique (BFR) can be seen as a promising alternative for promoting greater mechanical and muscular stress, thus providing a more efficient warm-up and optimizing performance. Objectives: to analyze the effects of RFS used during low-intensity warm-up compared with low-intensity and high-intensity warm-up without RFS on performance (jump test and 30-meter sprint test) and skin surface temperature. In addition to analyzing and comparing, after the warm-up protocols with and without RFS, the acute responses on perceptual outcomes (perception of pain, change in sensitivity, subjective perception of exertion and perception of discomfort in relation to RFS) and muscle outcomes (tonus , muscle stiffness and elasticity). Methods: a randomized controlled clinical trial will be carried out, with 33 amateur soccer players aged between 18 and 35 years who will be randomly divided into three groups: low-intensity warm-up without RFS (30% VO2max), high-intensity warm-up without RFS ( 80% VO2max) and low-intensity warm-up associated with BFR (80% of total occlusion pressure) [30% VO2max-BFR]. All groups will carry out the heating protocol and the outcomes will be evaluated at baseline and immediately after the end of the heating, as well as 10 and 20 minutes after its completion, namely: skin surface temperature through thermography; tone, stiffness and muscle elasticity by myotometry, subjective perception of pain (VAS); pain threshold through the pressure algometer; subjective perception of exertion (BORG scale); perception of discomfort in relation to RFS (LIKERT-CR-10 scale); 30-meter sprints measured through photocells and vertical jump, measured through the force platform. Descriptive statistics will be used and comparisons will be made using the generalized linear mixed model, assuming a significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* male
* healthy
* amateur soccer player
* aged between 18 and 35 years

Exclusion Criteria:

* smokers;
* alcoholics;
* use drugs that influenced cardiac autonomic activity;
* cardiovascular, metabolic or endocrine diseases;
* having one or more predisposing risk factors for thromboembolism;
* history of lower extremity surgery or musculoskeletal injury within the last six months that may impair your performance during testing or warm-up (e.g., meniscal repair, ligament reconstruction, muscle injury, tendinopathy, lower extremity patellofemoral pain, and/or back pain);

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Temperature | At the baseline
  Skin surface temperature will be evaluated using a thermographic camera
Temperature | Immediately after warm-up
  Skin surface temperature will be evaluated using a thermographic camera
Performance in Squat Jump Test | At the baseline
  The squat jump test will be performed at jumping platform (Multisprint, Hidrofit, Brazil)
Performance in Squat Jump Test | Immediately after warm-up
  The squat jump test will be performed at jumping platform (Multisprint, Hidrofit, Brazil)
Performance in 30 meter sprint | At the baseline
  the sprint test will be performed in a hall and two pairs of photoelectric cells (Multisprint®, Hidrofit, Brazil) will be used with an accuracy of 0.01 seconds.
Performance in 30 meter sprint | Immediately after warm-up
  the sprint test will be performed in a hall and two pairs of photoelectric cells (Multisprint®, Hidrofit, Brazil) will be used with an accuracy of 0.01 seconds.

SECONDARY OUTCOMES:
Pain threshold | At the baseline
  To assess the pain threshold, the pressure algometer will be applied at 10 specific locations on the lower limb
Pain threshold | Immediately after warm-up
  To assess the pain threshold, the pressure algometer will be applied at 10 specific locations on the lower limb
Muscle Pain | At the baseline
  The subjective evaluation of pain will be obtained through the Visual Analogue Scale (VAS), graded from 0 to 10, with zero being the total absence of pain and 10 the maximum level of pain supported by the participan
Muscle Pain | Immediately after warm-up
  The subjective evaluation of pain will be obtained through the Visual Analogue Scale (VAS), graded from 0 to 10, with zero being the total absence of pain and 10 the maximum level of pain supported by the participan
Perceived Effort Scale (Borg) | At the baseline and Immediately after warm-up
  The degree of subjective exertion reported by the participants in relation to the lower limbs will be analyzed by Borg's scale of perception of effort of 0 to 10 points, 0 being "very easy" and 10 being "exhaustive."
Perceived discomfort Scale (Likert-RFS) | At the baseline and Immediately after warm-up
  The degree of subjective discomfort reported by the participants in relation to the lower limbs refferd a blood flow restriction will be analyzed by Likert Scale of perception of effort of 0 to 10 points, 0 being "no discomfort" and 10 being "very discomfortable."
Resistance through Bioimpedance analysis (BIA) | At the baseline and Immediately after warm-up
  Evaluation of tissue resistance, the higher the value, the worse the result
Reactance through Bioimpedance analysis (BIA) | At the baseline and Immediately after warm-up
  Evaluation of tissue reactance, the higher the value, the better the cell integrity
Phase angle through Bioimpedance analysis (BIA) | At the baseline and Immediately after warm-up
  Assessment of the phase angle, the higher the value, the better the condition of the participant
Tone muscular through Myotonometry used the MyotonPRO equipment | At the baseline and Immediately after warm-up
  Natural Oscillation Frequency [Hz], characterizing Tone of the muscles: quadriceps femoris, biceps femoris, semitendinosus, triceps surae and tibialis anterior
Stiffness through Myotonometry used the MyotonPRO equipment | At the baseline and Immediately after warm-up
  Mechanical Stress Relaxation Time [ms] featuring muscle elasticity of the muscles: quadriceps femoris, biceps femoris, semitendinosus, triceps surae and tibialis anterior
heart rate variability indices in the time domain | At the baseline time (30 minutes rest in the supine position), during the warm-up (15 minutes in the treadmill) and immediately after the warm-up (60 minutes rest in the supine position)
  Mean RR, SDNN e rMSSD
heart rate variability indices in the frequency domain | At the baseline time (30 minutes rest in the supine position), during the warm-up (15 minutes in the treadmill) and immediately after the warm-up (60 minutes rest in the supine position)
  LF and HF in nu and ms2
heart rate variability indices analyzed in the Poincaré plot | At the baseline time (30 minutes rest in the supine position), during the warm-up (15 minutes in the treadmill) and immediately after the warm-up (60 minutes rest in the supine position)
  SD1 and SD2 in ms

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Carlos Alberto Toledo Teixeira Filho, Presidente Prudente, São Paulo
  - Franciele Marques Vanderlei, Presidente Prudente, São Paulo